CLINICAL TRIAL: NCT04033900
Title: Effect of Active Warming Prior to Surgery in Perioperative Hypothermia
Brief Title: Effects of Active Prewarming in Perioperative Hypothermia in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RECIO PÉREZ, JESÚS (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Sponsor-Investigator, RECIO PÉREZ, JESÚS, ANESTHESIOLOGIST, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200230
Record Dates: First submitted 2019-06-19; First posted 2019-07-26 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hypothermia; Anesthesia; Hypothermia Due to Anesthetic; Hypothermia Following Anesthesia; Hypothermia Following Anesthesia, Sequela
Keywords: Active preoperative warming; Inadvertent hypothermia; Perioperative hypothermia; Surgical prewarming; Forced air warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prewarming (Experimental): Active warming is allowed prior to surgery with forced-air warming devices
  Interventions: Device: Forced air warming devices
- No prewarming (No Intervention): Non active warming is allowed before surgery

INTERVENTIONS:
Device: Forced air warming devices — In the treatment group, heating will be started with a pre-surgical forced-air blanket "Outpatient Warming Blanket model 11101 Bair Hugger from 3M" and a forced-air heating unit "Bair Hugger Warming Unit Model 775 from 3M" at 38-43º C which will be maintain during the stay in the pre-surgery room until the transfer to the operating room
  Other Names: Outpatient Warming Blanket Model 11101 Bair Hugger 3M; BAir Hugger Warming Unit Model 775 3M
  Arms: Prewarming

SUMMARY:
This study evaluates the effect of active prewarming on the frequency and duration of perioperative hypothermia. 50% of patients will receive active warming with forced-air devices prior to entering the operating room, and the other 50% will not receive any active heating measures.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia is defined as a body temperature below 36º C during the perioperative period. It occurs as a result of the effects of anesthetic drugs on the regulation of body temperature and exposure to a cold environment.

The main temperature loss during the perioperative period occurs during the first hour after the anesthetic induction as a result of heat redistribution from the central compartment to the peripheral compartment

The most effective strategy to prevent perioperative hypothermia is the use of forced-air warming devices. These devices are usually initiated once the patient enters the operating room. At that time, the patient has already initiated the heat loss by distributing heat from the central to the peripheral compartment to maintain body temperature.

We intend to use forced-air warming devices before the patients is transferred to the operating room in order to preserve the peripheral body temperature. This way the redistribution of heat should be avoided and, therefore, perioperative hypothermia and its harmful effects will be prevented.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old.
* American Society of Anesthesiologists I-III.
* Undergoing surgery under general or locoregional anesthesia lasting more than 30 minutes.
* General surgery: hernias, cholecystectomies, hepatectomies, intestinal resections, pancreatoduodenectomies ...
* Traumatology and orthopedics: total / partial knee prosthesis, total / partial hip prosthesis, osteosynthesis, removal of material, arthroscopies, hallux valgus, lumbar arthrodesis ...
* Neurosurgery: lumbar arthrodesis, excision of intracranial tumors.
* Gynecology: Hysterectomies, adnexectomies, hysteroscopy ...
* Otorhinolaryngology: septoplasty, nasosinusal endoscopic surgery, tonsillectomies, adenoidectomies, thyroidectomies...
* Thoracic: Pneumonectomies and pulmonary resections, sympathectomies, thoracoscopy ...
* Urology: Bladder transurethral resection , prostate transurethral resection, nephrectomies.
* Maxillofacial: parathyroidectomies, microsurgery ...
* Ability to understand the study, give authorization and collaborate with data collection

Exclusion Criteria:

* Local anesthesia or peripheral nerve block.
* Urgent or emergent surgery.
* Cognitive impairment or lack of collaboration of any kind
* Pregnant women undergoing cesarean section.
* Diabetes Mellitus poorly controlled (HbA1c> 6.5-7%)
* Subjects that are under treatment with drugs that interfere with thermoregulation or may cause drug-induced hyperthermia (amphetamines, barbiturates, inhaled gases ...)
* Subjects with burns, pressure ulcers and other surface disturbances that cover the heating devices
* Subjects with screening temperature > 37.5º C.
* Subjects with fever or active infections.
* Subjects with chronic anemia who require periodic transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative hypothermia | From 1 hour to 12 hours
  Core temperature below 36º C measured with 3M Spot On monitor every 5 minutes from arrival to the pre-surgical area, during surgery and unit discharge to the ward

SECONDARY OUTCOMES:
Hypothermia duration | Minutes with core temperature below 36ºC from arrival to the OR unit discharge to postoperative unit, up to 10 hours, whichever came first.
  Time of core temperature below 36º C measured every 5 minutes with 3M Spot On monitor from arrival to the surgery room and unit discharge to postoperative unit.
Hospital stay | From date of Admission in hospital until the date of discharge from hospital, assessed up to 120 days.
  Patient´s days keep in hospital, from admission in hospital until discharge from the home
Surgical site infection | 1 Month
  Follow-up the wound and evaluation of signs and symptoms of surgical site infection from surgery to review for the nurse.
Prewarming duration | From 10 minutes to 1 hour
  Time from pre-warming initiation in pre operative area with forced air warming device until transfer to operating theatre.

CONTACTS AND LOCATIONS:
Overall Officials: JESÚS RECIO PÉREZ, ANESTHETIST, Principal Investigator — HOSPITAL UNIVERSITARIO DE TORREJON
Locations (1):
- Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid, Spain

REFERENCES:
- [Background] Warttig S, Alderson P, Campbell G, Smith AF. Interventions for treating inadvertent postoperative hypothermia. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD009892. doi: 10.1002/14651858.CD009892.pub2. PMID 25411963
- [Background] Giuliano KK, Hendricks J. Inadvertent Perioperative Hypothermia: Current Nursing Knowledge. AORN J. 2017 May;105(5):453-463. doi: 10.1016/j.aorn.2017.03.003. PMID 28454611
- [Background] Madrid E, Urrutia G, Roque i Figuls M, Pardo-Hernandez H, Campos JM, Paniagua P, Maestre L, Alonso-Coello P. Active body surface warming systems for preventing complications caused by inadvertent perioperative hypothermia in adults. Cochrane Database Syst Rev. 2016 Apr 21;4(4):CD009016. doi: 10.1002/14651858.CD009016.pub2. PMID 27098439
- [Background] Torossian A, Brauer A, Hocker J, Bein B, Wulf H, Horn EP. Preventing inadvertent perioperative hypothermia. Dtsch Arztebl Int. 2015 Mar 6;112(10):166-72. doi: 10.3238/arztebl.2015.0166. PMID 25837741
- [Background] Wagner D, Byrne M, Kolcaba K. Effects of comfort warming on preoperative patients. AORN J. 2006 Sep;84(3):427-48. doi: 10.1016/s0001-2092(06)63920-3. PMID 17004666
- [Background] Kellam MD, Dieckmann LS, Austin PN. Forced-air warming devices and the risk of surgical site infections. AORN J. 2013 Oct;98(4):354-66; quiz 367-9. doi: 10.1016/j.aorn.2013.08.001. PMID 24075332
- [Background] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088